CLINICAL TRIAL: NCT01280565
Title: A Prospective, Multicenter, Randomized, Open-label, Active Controlled, Two-parallel Groups, Phase 3 Study to Compare the Efficacy and Safety of Masitinib at 7.5 mg/kg/Day to Dacarbazine in the Treatment of Patients With Non-resectable or Metastatic Stage 3 or Stage 4 Melanoma Carrying a Mutation in the Juxta Membrane Domain of C-kit
Brief Title: Masitinib in Non-Resectable or Metastatic Stage 3/4 Melanoma Carrying a Mutation in the Juxta Membrane Domain of c-Kit
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB08026
Record Dates: First submitted 2010-08-06; First posted 2011-01-21 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Tyrosine kinase inhibitor; c-Kit juxta membrane mutation
MeSH Terms: conditions — Melanoma | interventions — masitinib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Masitinib (Experimental): Participants receive masitinib (7.5 mg/kg/day), given orally twice daily.
  Interventions: Drug: Masitinib
- Dacarbazine (Active Comparator): Participants receive dacarbazine, given via IV bolus at 1,000 mg/m2 once every 3 weeks. Following a protocol amendment, the dacarbarzine treatment group has been closed
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: Masitinib — Masitinib 7.5 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib
Drug: Dacarbazine — IV bolus at 1,000 mg/m2 once every 3 weeks
  Other Names: DTIC
  Arms: Dacarbazine

SUMMARY:
The objective is to assess the efficacy and safety of masitinib at 7.5 mg/kg/day in the treatment of patients with non-resectable or metastatic stage 3 or stage 4 melanoma carrying a mutation in the juxta membrane domain of c-Kit and who have not previously been treated for melanoma.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor with potent activity against the juxta membrane domain of c-Kit. Masitinib is also thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective of this study was to evaluate the efficacy and safety of masitinib with respect to dacarbazine in the treatment of non-resectable or metastatic stage 3 or stage 4 melanoma carrying a mutation in the juxta membrane domain of c-Kit. Following a protocol amendment, the dacarbarzine treatment group was closed and recruitment restricted to masitinib treatment of chemo-naïve (first-line) patients.

ELIGIBILITY:
Main inclusion criteria include:

* Patient with histologically or cytologically confirmed non-resectable or metastatic stage 3 (non-resectable IIIB or IIIC, AJCC TNM staging system 7th edition) or stage 4 melanoma
* Patient with detectable c-Kit JM mutation (mutation in exon 9, 11 or 13) confirmed by DNA or RNA sequencing, which is expected to be mainly found after screening of mucosal or acral melanoma or melanoma on skin with chronic sun-induced damages (defined by a microscopically marked elastosis involving the skin surrounding their primary melanoma).
* Patient not previously treated for melanoma (first-line)

Main exclusion criteria include:

* Pregnant, or nursing female patient
* Patient with active brain metastases.
* Prior treatment with a tyrosine kinase c-Kit inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 24 weeks
  Estimated as the number of patients with documented partial response or complete response defined according to the RECIST criteria, divided by the number of randomized patients

SECONDARY OUTCOMES:
PFS | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival (PFS) is defined as the delay between the date of randomization to the date of documented progression (according to RECIST) or any cause of death during the study.
Overall Survival (OS) | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques GROB, MD, PhD, Principal Investigator — Hôpital Sainte Marguerite, Marseille, France
Locations (9):
- Blumenthal Cancer Centre, Charlotte, North Carolina, United States
- University Hospital Hradec Králové, Hradec Králové, Czechia
- France (3):
  - Hôpital Saint Andre, Bordeaux
  - Centre Hospitalier LE MANS, Le Mans
  - Hôpital Sainte Marguerite, Marseille
- Klinik und Poliklinik für Hautkrankheiten, Münster, Germany
- Istituto Europeo di Oncologia, Milan, Italy
- N.N.Blokhin Russian Cancer Research Centre, Moscow, Russia
- Hospital General de Valencia, Valencia, Spain